CLINICAL TRIAL: NCT05179577
Title: A Randomized, Double-Blind, Placebo-Controlled Parallel Group Study to Investigate the Safety and Efficacy of Arbaclofen Extended-Release Tablets for the Treatment of Spasticity in Patients With Multiple Sclerosis (Study OS440-3006)
Brief Title: A Study to Investigate Arbaclofen ER Tablets for the Treatment of Spasticity in Patients With Multiple Sclerosis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RVL Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OS440-3006
Record Dates: First submitted 2021-11-12; First posted 2022-01-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Spasticity
MeSH Terms: conditions — Muscle Spasticity | interventions — arbaclofen placarbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arbaclofen Extended-Release (Active Comparator): Extended-release oral tablet, twice daily dosing (80 mg/day)
  Interventions: Drug: Arbaclofen
- Placebo (Placebo Comparator): Extended-release oral tablet, twice daily dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arbaclofen — Arbaclofen Extended Release Tablets
  Other Names: OS440; AERT
  Arms: Arbaclofen Extended-Release
Drug: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the safety and efficacy of oral arbaclofen ER tablets in MS patients with spasticity. Arbaclofen ER will be compared with placebo.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the safety and efficacy of oral arbaclofen ER tablets (80 mg/day) in MS patients with spasticity. Arbaclofen ER will be compared with placebo. The treatment groups will be randomized in a 1:1 ratio. There will be a 49-day dose escalation period, followed by a 84-day maintenance treatment period, followed by a 21-day taper period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 to 65 years of age, inclusive
* An established diagnosis per McDonald Criteria (Polman et al 2011) of MS (either RR or SP course) that manifests a documented history of spasticity for at least 6 months prior to screening
* Spasticity due to MS as shown by a TNmAS-MAL score ≥ 2
* Expanded Disability Status Scale (EDSS) score greater than or equal to (≥) 3.0 and less than or equal to (≤) 7.0
* Absence of infections, peripheral vascular disease, painful contractures, advanced arthritis, or other conditions that hinder evaluation of joint movement
* Use of a medically highly effective form of birth control (see Section 7.8) during the study and for 3 months thereafter for women of child-bearing potential (including female subjects and female partners of non-sterile male subjects)
* Willing to sign the informed consent form (ICF)

Exclusion Criteria:

* Any concomitant disease or disorder that has symptoms of spasticity or that may influence the subject's level of spasticity
* In the opinion of the investigator, the patient is unable to rate their level of spasticity or distinguish it from other MS symptoms
* Concomitant use of medications that would potentially interfere with the actions of the study medication or outcome variables
* Pregnancy, lactation, or planned pregnancy during the course of the study and for 3 months after the final study visit
* Current significant cognitive deficit, severe or untreated anxiety, severe or untreated depression
* Current malignancy or history of malignancy that has not been in remission for more than 5 years, except effectively treated basal cell skin carcinoma
* Any other significant disease, disorder, or significant laboratory finding which, in the opinion of the investigator, puts the subject at risk because of participation, influences the result of the study, or affects the subject's ability to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Maintenance Treatment Period for Total Numeric-Transformed Modified Ashworth Scale Most Affected Limb (TNmAS-MAL) | Maintenance Treatment Period: Visit 5 (day 77), Visit 6 (day 105), and Visit 7 (day 133)
  The total numerical score of a limb accounts for the sum of the 3 main joint muscular group scores. The limb with the highest score is the most affected limb. Lower score is better. Scale is from 0 to 5.
Responder Analysis of Ashworth Scale Score (AS-MAL-R) for Maintenance Treatment Period | Maintenance Treatment Period: Visit 5 (day 77), Visit 6 (day 105), and Visit 7 (day 133)
  Responder status (AS-MAL-R) consists of three response categorical outcomes based on the Ashworth Scale (AS). Where the possible outcomes are: Strong Responder, Responder, or Non-Responder

SECONDARY OUTCOMES:
Change from Baseline to Maintenance Treatment Period for Total Numeric-Transformed Modified Ashworth Scale Total Limbs (TNmAS-TL) | Maintenance Treatment Period: Visit 5 (day 77), Visit 6 (day 105), and Visit 7 (day 133)
  The total numerical score of a limb accounts for the sum of the 3 main joint muscular group scores. The total of the 4 limbs is the total limbs score. Lower score is better. Scale is from 0 to 5 per joint, Maximum score per limb is 15. Maximum total limbs score is 60.
Clinician's global impression of change (CGIC) for Maintenance Treatment Period | Maintenance Treatment Period: Visit 5 (day 77), Visit 6 (day 105), and Visit 7 (day 133)
  The clinician makes a judgment about the change from baseline of illness severity, the subject's level of distress, other aspects of impairment, and the impact of the illness on functioning. Scale of -3 to +3, higher score is better
Numeric Rating Scale of Spasticity (NRS-S) for Maintenance Treatment Period | Maintenance Treatment Period: Visit 5 (day 77), Visit 6 (day 105), and Visit 7 (day 133)
  The Numeric Rating Scale of Spasticity is a patient rated measure of the perceived severity of spasticity using a 0-10 numeric rating scale. Lower score is better.
Expanded Disability Status Scale (EDSS) for Maintenance Treatment Period | Maintenance Treatment Period: Visit 5 (day 77), Visit 6 (day 105), and Visit 7 (day 133)
  EDSS is a method of quantifying disability in MS and monitoring changes in the level of disability over time. Scale ranges from 0-10, in 0.5 unit increments. Lower score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Tina deVries, PhD, Study Director — RVL Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No